CLINICAL TRIAL: NCT00847873
Title: Treatment of Intimate Partner Violence and Substance Abuse in a Substance Abuse: a Randomized Controlled Trial
Brief Title: Treatment of Intimate Partner Violence and Substance Abuse in a Substance Abuse Treatment Facility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Paul M.G.Emmelkamp, Prof. Dr. P.M.G. Emmelkamp, VU University of Amsterdam
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2008-KP-466
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Domestic Violence; Substance Abuse
Keywords: intimate partner violence; domestic violence; alcohol abuse; alcohol dependence; drug abuse; drug dependence; addiction
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism; Behavior, Addictive | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combined SU/IPV treatment (Experimental): A combined treatment containing cognitive behavioral therapy addressing partner violence and cognitive behavioral therapy addressing substance abuse
  Interventions: Behavioral: substance abuse/domestic violence treatment
- control condition (Active Comparator): Cognitive behavioral therapy addressing substance abuse
  Interventions: Behavioral: Cognitive behavioral therapy addressing substance abuse

INTERVENTIONS:
Behavioral: substance abuse/domestic violence treatment — This intervention is comprised of 16 sessions of cognitive behavioral therapy. 8 sessions are addressing partner violence and 8 sessions are addressing substance abuse
  Other Names: Treatment for intimate partner violence; Treatment for addiction
  Arms: Combined SU/IPV treatment
Behavioral: Cognitive behavioral therapy addressing substance abuse — This intervention is comprised of 16 sessions of cognitive behavioral therapy addressing substance abuse.
  Other Names: Treatment for addiction
  Arms: control condition

SUMMARY:
Intimate partner violence is a significant societal problem. There is considerable evidence that a strong relationship between the use of alcohol and other drugs and intimate partner violence exists. Besides, a few studies indicate that reducing substance use may have a positive impact on IPV. Therefore, in this study, patients in substance abuse treatment for the use of alcohol, cannabis or cocaine who also admit to perpetrating intimate partner violence will be randomly assigned to either cognitive behavioral therapy addressing substance abuse combined with treatment for offenders of intimate partner violence or substance abuse treatment alone.

DETAILED DESCRIPTION:
Intimate partner violence is a significant societal problem. However, treatment of IPV perpetrators is far from effective, which may be partly due to the fact that the role of substance abuse is not taken into account. There is considerable evidence that a strong relationship between the use of alcohol and other drugs and intimate partner violence exists. Besides, a few studies indicate that reducing substance use may have a positive impact on IPV. Therefore, in this study, patients in substance abuse treatment for the use of alcohol, cannabis or cocaine who also admit to perpetrating intimate partner violence will be randomly assigned to either cognitive behavioral therapy addressing substance abuse combined with treatment for offenders of intimate partner violence or substance abuse treatment alone.

ELIGIBILITY:
Inclusion Criteria:

* Perpetration of intimate partner violence in the past year
* Substance abuse or dependence (current)
* Currently in a relationship

Exclusion Criteria:

* Not sufficient fluency in Dutch to complete treatment and measures
* (Ab)use of crack cocaine and/or heroin
* Psychosis
* Psychopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-10; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Substance use: Timeline followback interview (TLFB) | pretest, posttest, 6 & 12 months follow-up
IPV: Conflict Tactics Scale 2 (CTS2) | pretest, halfway treatment, posttest, 6 and 12 months follow-up

SECONDARY OUTCOMES:
Brief Symptom Inventory (BSI) | pretest, posttest
Substance use: Quick drinking and drug use screen | Pretest, halfway treatment, posttest, 6 and 12 months follow-up
Maudsley Marital Questionnaire (MMQ) | Pretest, posttest, 6 and 12 months follow-up
Treatment Satisfaction Questionnaire | posttest

CONTACTS AND LOCATIONS:
Overall Officials: Paul M. Emmelkamp, PhD., Principal Investigator — University of Amsterdam
Locations (1):
- JellinekMentrum, Amsterdam, Netherlands